CLINICAL TRIAL: NCT01935193
Title: Impact of Different Pharmacological Formulations on Aspirin Resistance Reversibility in Diabetics Patients
Brief Title: Aspirin Resistance Reversibility in Diabetic Patients
Acronym: ARRDM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Responsible Party: Principal Investigator, Marta Bisi, MD, Azienda Ospedaliera San Giovanni Battista
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASAR160
Record Dates: First submitted 2013-08-28; First posted 2013-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-08

CONDITIONS: Aspirin Resistance
Keywords: platelets aggregation; asa resistance
MeSH Terms: interventions — acetylsalicylic acid lysinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- asa resistant (Experimental): asa resistant patients receive endovenous infusion of lysine acetylsalicylate 288 mg and if asa resistance has been reversed they have been prescribed oral soluble salt of lysine acetylsalicylate.
  Interventions: Drug: lysine acetylsalicylate

INTERVENTIONS:
Drug: lysine acetylsalicylate
  Other Names: Flectadol; Cardirene

SUMMARY:
The aim of the study is assessing the prevalence of aspirin resistance in a cohort of diabetic patients. Those found resistant has been undergone pharmacological tests using different drug formulations to investigate the reversibility of aspirin resistance.

ELIGIBILITY:
Inclusion Criteria:

* diabete mellitus type 2
* asa since 30 days at least
* plts >150000 and <450000

Exclusion Criteria:

* recent ACS (within 30 days)
* anticoagulant therapy
* haemorragic diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
platelets aggregation assessed by two tests (PFA100 and VerifyNow) | 24 hours
  diabetic patients found aspirin resistant receive and infusion of 288 mg of lysine acetylsalicylate and they are tested again 24 h after the infusion to investigate if aspirin resistance have been reversed.

SECONDARY OUTCOMES:
stability of aggregation state after the reversion of aspirin resistance using oral formulation of lysine acetylsalicylate | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- San Giovanni Battista Hospital, Torino, Italy